CLINICAL TRIAL: NCT02406053
Title: Evaluation of Oxidative Damage and Antioxidant Mechanisms in COPD, Lung Cancer, and Obstructive Sleep Apnea Syndrome
Brief Title: Oxidative Damage and Antioxidant Mechanisms in COPD
Status: Completed | Type: Observational
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Aysel Sünnetçioğlu, Department of Pulmory Diseas Aysel Sünnetçioğlu, Yuzuncu Yil University
Other Study IDs: YYU-016; YYU-2015-66 (Other: YUZUNCU YIL UNIVERSITY)
Record Dates: First submitted 2015-03-16; First posted 2015-04-02 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Respiratory Diseases
Keywords: lung cancer; antioxidants; oxidative damage
MeSH Terms: conditions — Respiratory Tract Diseases; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- OSAS: Obstructive sleep apnea syndrome
  Interventions: Genetic: oxidative and antioxidant biomarkers
- COPD: Chronic obstructive pulmonary disease
  Interventions: Genetic: oxidative and antioxidant biomarkers
- LC: Lung cancer
  Interventions: Genetic: oxidative and antioxidant biomarkers
- HC: Healthy controls
  Interventions: Genetic: oxidative and antioxidant biomarkers

INTERVENTIONS:
Genetic: oxidative and antioxidant biomarkers — the oxidative damage in these diseases by evaluating the oxidative and antioxidant biomarkers.

SUMMARY:
The environmental pollutants and endogenous reactive oxygen metabolites from inflammatory cells exert substantial pathological effects on the lung cells [1]. Oxidative stress (OS) is a major factor that plays a significant role in lung cancer (LC) [2], chronic obstructive pulmonary disease (COPD) [3] and obstructive sleep apnea syndrome (OSAS) [4, 5]. The current evidence suggests that OS takes part in the mechanisms involved in initiation, promotion and progression of respiratory diseases. The major exposures that cause OS can be summarized as smoking, and ambient air pollution that contains particulate matter smaller than aerodynamic diameter of 2.5 µm [6-8]. Epidemiological and clinical studies showed that the overall outcome of pulmonary OS is increased mortality due to increased incidence of respiratory diseases [9].

DETAILED DESCRIPTION:
Introduction Lung is a particularly important organ because of its interface with the environment. The environmental pollutants and endogenous reactive oxygen metabolites from inflammatory cells exert substantial pathological effects on the lung cells [1]. Oxidative stress (OS) is a major factor that plays a significant role in lung cancer (LC) [2], chronic obstructive pulmonary disease (COPD) [3] and obstructive sleep apnea syndrome (OSAS) [4, 5]. The current evidence suggests that OS takes part in the mechanisms involved in initiation, promotion and progression of respiratory diseases. The major exposures that cause OS can be summarized as smoking, and ambient air pollution that contains particulate matter smaller than aerodynamic diameter of 2.5 µm [6-8]. Epidemiological and clinical studies showed that the overall outcome of pulmonary OS is increased mortality due to increased incidence of respiratory diseases [9].

In OSAS, an episodic hypoxia-reoxygenation cycle occurs during intermittent nocturnal hypoxias that causes the production of reactive oxygen metabolites [10]. These metabolites are responsible for the activation of inflammatory cells in OSAS [11, 12], and their increased levels eventually cause ischemia-reperfusion injury [13], and cellular and DNA damage [14, 15]. The latter, is also a significant contributor of LC progression. The DNA damage in the presence of reactive oxygen metabolites yields carcinogenesis by several mechanisms. Some of them are single or double-stranded DNA breaks, and modifications in purines or pyrimidines. Nevertheless, OS is not the only susceptible factor for carcinogenesis, there are also many other pathological mechanisms contributing to cancer development, such as reactive nitrogen species, and involvement of mitochondrial DNA mutations [16] in inflammatory conditions. Previous studies reported that LC occurs two-to-five times higher in patients with moderate-to-severe COPD [17, 18]. OS is also the main etiological factor of COPD, which is particularly important in the acute exacerbations of the disease [19]. The parenchymal damage in COPD includes some mechanisms such as chronic inflammation, OS, deteriorations in the balance of protease and antiprotease activities, and apoptosis [20]. The major etiological factor that suspected to play role in the progression of LC in COPD is reported as chronic inflammation, which causes induction of several interleukins and cyclooxygenase-2 activity. The inflammatory micro-environment is a potential medium for contributing the neoproliferative process, which interacts with regulatory mechanism such as apoptosis and angiogenesis [21].

Some biomarkers are available for evaluating the OS in the living organisms [22]. Some of these biomarkers are malondialdehyde (MDA), 8-oxo-7,8-dihydro-2'-deoxyguanosine (8-OHdG), and coenzyme Q10 (CoQ10). Each of these biomarkers is involved in oxidative processes. MDA is a by-product of polyunsaturated fatty acid peroxidation [23]. Lipid peroxidation is the oxidation reactions between reactive oxygen metabolites and polyunsaturated fatty acids, which eventually causes changes in the structure and permeability of lung membrane [24]. The second biomarker, 8-OHdG, is primarily involved in DNA damage. The mechanism for this damage is the guanine: cytosine to adenine: thymine transversion on DNA replication [25], which induces microsatellite instability, and abnormal apoptosis or necrosis [26]. The third biomarker is CoQ10, which is also a mediator of lipid peroxidation, and an essential cofactor in the electron-transport chain (ETC). It is also a lipophilic antioxidant component of the lipid membranes [27]. In this study.

ELIGIBILITY:
Inclusion Criteria:

* Malondialdehyde (MDA), 8-oxo-7,8-dihydro-2'-deoxyguanosine (8-OHdG), and coenzyme Q10 (CoQ10) levels were evaluated in the blood samples of patients with COPD, LC, and OSAS by high-pressure liquid chromatography method.

Exclusion Criteria:

* The diagnosis of lung cancer was based on the analysis of biopsy or cytologic specimens obtained by bronchoscopic examination, transthoracic biopsy or surgery. The patients Who hadn't have chemo or/and radiotherapy were included to the study.
* The exclusion criteria for COPD, OSAS and lung cancer were the presence of the following: history of cardiovascular disease, hypertension, diabetes mellitus, inﬂammatory or infectious.

Ages: 38 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 111 participants (35 females, 76 males) with OSAS (n=29), COPD (n=26) and LC (n=28), and healthy controls (n=28) were included in the study.
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Oxidative damage by evaluating the oxidative and antioxidant biomarkers | 4 months
  This study aimed to evaluate the oxidative damage in these diseases by evaluating the oxidative and antioxidant biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: AYSEL SUNNETCIOGLU, Phd, Principal Investigator — Yuzuncu Yil University

REFERENCES:
- [Derived] Sunnetcioglu A, Alp HH, Sertogullarindan B, Balaharoglu R, Gunbatar H. Evaluation of Oxidative Damage and Antioxidant Mechanisms in COPD, Lung Cancer, and Obstructive Sleep Apnea Syndrome. Respir Care. 2016 Feb;61(2):205-11. doi: 10.4187/respcare.04209. Epub 2015 Nov 24. PMID 26604330